CLINICAL TRIAL: NCT01209286
Title: An Open Label, Multicenter, Exploratory Phase II Study to Evaluate the Efficacy, Safety, and Tolerability of the BiTE® Antibody Blinatumomab in Adult Patients With Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia (ALL)
Brief Title: Study of the BiTE® Blinatumomab (MT103) in Adult Patients With Relapsed/Refractory B-Precursor Acute Lymphoblastic Leukemia (ALL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen Research (Munich) GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT103-206
Record Dates: First submitted 2010-09-23; First posted 2010-09-27 (Estimated); Results first posted 2015-01-07 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2016-07

CONDITIONS: B-ALL
Keywords: Blinatumomab; B-ALL; adult ALL; relapsed ALL; refractory ALL; Leukemia; ALL; Lymphatic diseases; Lymphoproliferative disorders; bispecific antibody; anti-CD19; Immunotherapeutic treatment
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Lymphatic Diseases; Lymphoproliferative Disorders | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Blinatumomab 15 μg (Experimental): Participants received blinatumomab 15 μg/m²/day as a continuous intravenous infusion at a constant flow rate over 4 weeks followed by a 2-week treatment-free interval for up to 5 consecutive cycles.
  Interventions: Biological: Blinatumomab
- Blinatumomab 5/15 μg (Experimental): Participants received blinatumomab by continuous intravenous infusion over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. The initial dose was 5 μg/m²/day for the first seven days of treatment, followed by 15 μg/m²/day starting from Week 2 of treatment.
  Interventions: Biological: Blinatumomab
- Blinatumomab 5/15/30 μg (Experimental): Participants received blinatumomab by continuous intravenous infusion over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. The initial dose was 5 μg/m²/day for the first seven days of treatment, a dose of 15 μg/m²/day in the subsequent 7 days, followed by 30 μg/m²/day starting from Week 3 of treatment.
  Interventions: Biological: Blinatumomab

INTERVENTIONS:
Biological: Blinatumomab — Continuous intravenous infusion over four weeks per treatment cycle
  Other Names: AMG103; MT103; BLINCYTO™

SUMMARY:
The purpose of this study is to determine whether the bispecific T-cell engager blinatumomab is effective, safe and tolerable in the treatment of patients with relapsed/refractory B-precursor ALL.

DETAILED DESCRIPTION:
Relapsed/refractory B-precursor ALL in adult patients is an aggressive malignant disease with dismal prognosis and unmet medical need. Additional therapeutic approaches are urgently needed. Blinatumomab is a bispecific single-chain antibody construct designed to link B cells and T cells resulting in T cell activation and a cytotoxic T cell response against CD19 expressing cells. The purpose of this study is to investigate the efficacy, safety and tolerability of different doses of the bispecific T-cell engager blinatumomab in adult patients with relapsed/refractory B-precursor ALL. Patrticipants will receive up to five 4-week cycles of intravenous blinatumomab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with B-precursor ALL relapsed after at least induction and consolidation or having refractory disease
* More than 5% blasts in bone marrow
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Life expectancy of ≥ 12 weeks

Exclusion Criteria:

* History or presence of clinically relevant central nervous system (CNS) pathology
* Infiltration of cerebrospinal fluid (CSF) by ALL
* Autologous/allogeneic hematopoietic stem cell transplantation (HSCT) within six weeks/three months prior to start of blinatumomab treatment
* Active Graft-versus-Host Disease (GvHD)
* Patients with Philadelphia chromosome (Ph)+ ALL eligible for treatment with dasatinib or imatinib
* Cancer chemotherapy within two weeks prior to start of blinatumomab treatment
* Immunotherapy (e.g. rituximab) within four weeks prior to start of blinatumomab treatment
* Infection with human immunodeficiency virus (HIV) or hepatitis B (HBsAg positive) or hepatitis C virus (anti-HCV positive)
* Pregnant or nursing women
* Previous treatment with blinatumomab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-10; Primary Completion 2012-03 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Max Topp, MD, Principal Investigator — University of Wuerzburg
Locations (9):
- Germany (9):
  - Frankfurt
  - Freiburg im Breisgau
  - Hanover
  - Kiel
  - Münster
  - Regensburg
  - Tübingen
  - Ulm
  - Würzburg

REFERENCES:
- [Derived] Nagele V, Kratzer A, Zugmaier G, Holland C, Hijazi Y, Topp MS, Gokbuget N, Baeuerle PA, Kufer P, Wolf A, Klinger M. Changes in clinical laboratory parameters and pharmacodynamic markers in response to blinatumomab treatment of patients with relapsed/refractory ALL. Exp Hematol Oncol. 2017 May 18;6:14. doi: 10.1186/s40164-017-0074-5. eCollection 2017. PMID 28533941
- [Derived] Zhu M, Wu B, Brandl C, Johnson J, Wolf A, Chow A, Doshi S. Blinatumomab, a Bispecific T-cell Engager (BiTE((R))) for CD-19 Targeted Cancer Immunotherapy: Clinical Pharmacology and Its Implications. Clin Pharmacokinet. 2016 Oct;55(10):1271-1288. doi: 10.1007/s40262-016-0405-4. PMID 27209293
- [Derived] Topp MS, Gokbuget N, Zugmaier G, Klappers P, Stelljes M, Neumann S, Viardot A, Marks R, Diedrich H, Faul C, Reichle A, Horst HA, Bruggemann M, Wessiepe D, Holland C, Alekar S, Mergen N, Einsele H, Hoelzer D, Bargou RC. Phase II trial of the anti-CD19 bispecific T cell-engager blinatumomab shows hematologic and molecular remissions in patients with relapsed or refractory B-precursor acute lymphoblastic leukemia. J Clin Oncol. 2014 Dec 20;32(36):4134-40. doi: 10.1200/JCO.2014.56.3247. Epub 2014 Nov 10. PMID 25385737

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was open to adult patients with relapsed / refractory B-precursor acute lymphoblastic leukemia (ALL).
Pre-assignment Details: This ongoing study consisted of a core study of up to 33 weeks, efficacy follow-up until 24 months after treatment start and survival follow-up until 5 years after treatment start. Data are reported for the primary analysis conducted when the last participant completed the core study; data cutoff date of 15 October 2012.
Period: Overall Study
Arm/Group | Blinatumomab 15 μg | Blinatumomab 5/15 μg | Blinatumomab 5/15/30 μg
Started | 7 | 23 | 6
Completed | 2 | 13 | 3
Not Completed | 5 | 10 | 3
Not completed — Adverse Event | 4 | 3 | 1
Not completed — Hematological Relapse After Remission | 0 | 1 | 1
Not completed — Remission Not Achieved in 2 Cycles | 1 | 3 | 1
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blinatumomab 15 μg | Blinatumomab 5/15 μg | Blinatumomab 5/15/30 μg | Total
Number analyzed (Participants) | 7 | 23 | 6 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (21.5) | 38.1 (16.7) | 42.5 (23.2) | 40.0 (18.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 2 | 14
  Male | 4 | 14 | 4 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 22 | 6 | 35
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Number of Prior Relapses [Number; unit: participants]
  0 | 0 | 2 | 1 | 3
  1 | 5 | 15 | 3 | 23
  2 | 2 | 6 | 1 | 9
  3 | 0 | 0 | 1 | 1
Relapsed / refractory Status [Number; unit: participants]
  Primary Refractory | 0 | 2 | 1 | 3
  Relapsed | 7 | 21 | 5 | 33
Prior Allogeneic Hematopoietic Stem cell Transplantation (HSCT) [Number; unit: participants]
  Yes, Sibling | 1 | 1 | 1 | 3
  Yes, Unrelated | 2 | 9 | 1 | 12
  Yes, Haploidentical (mother/father) | 0 | 0 | 0 | 0
  No prior allogeneic HSCT | 4 | 13 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Best Response of Complete Remission or Complete Remission With Only Partial Hematological Recovery Within 2 Cycles of Treatment
Description: At the end of each infusion period, a bone marrow aspiration/biopsy was performed to evaluate the efficacy of blinatumomab. All hematological assessments of bone marrow were reviewed in a central reference laboratory. Hematological remissions were defined by the following criteria:
  Complete Response/Remission (CR):
  * Less than or equal to 5% blasts in the bone marrow
  * No evidence of circulating blasts or extramedullar disease
  * Full recovery of peripheral blood counts:
    * Platelets > 100,000/μL
    * Hemoglobin ≥ 11 g/dL
    * Absolute neutrophil count (ANC) > 1,500/μL
  Complete Remission with only Partial Hematological Recovery (CRh*):
  * Less than or equal to 5% blasts in the bone marrow
  * No evidence of circulating blasts or extramedullar disease
  * Partial recovery of peripheral blood counts:
    * Platelets > 50,000/μL
    * Hemoglobin ≥ 7 g/dL
    * ANC > 500/μL.
Time Frame: Within the first 2 cycles of treatment, 12 weeks
Population: Full analysis set (FAS), defined as participants who received any infusion of the assigned study medication, who completed at least the first treatment cycle and for whom at least one response assessment was available after the start of treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Blinatumomab Overall: Participants received blinatumomab as a continuous intravenous infusion at a constant flow rate over 4 weeks followed by a 2-week treatment-free interval for up to 5 consecutive cycles.
Arm/Group | Blinatumomab 15 μg | Blinatumomab 5/15 μg | Blinatumomab 5/15/30 μg | Blinatumomab Overall
Number analyzed (Participants) | 7 | 23 | 6 | 36
percentage of participants | 71.4 [29.0 to 96.3] | 69.6 [47.1 to 86.8] | 66.7 [22.3 to 95.7] | 69.4 [51.9 to 83.7]

2. Secondary Outcome: Percentage of Participants With a Best Response of Complete Remission Within 2 Cycles of Treatment
Description: At the end of each infusion period, a bone marrow aspiration/biopsy was performed to evaluate the efficacy of blinatumomab. All hematological assessments of bone marrow were reviewed in a central reference laboratory. Complete Response/Remission (CR) was defined by the following criteria:
  * Less than or equal to 5% blasts in the bone marrow
  * No evidence of circulating blasts or extramedullar disease
  * Full recovery of peripheral blood counts:
    * Platelets > 100,000/μL
    * Hemoglobin ≥ 11 g/dL
    * Absolute neutrophil count (ANC) > 1,500/μL
Time Frame: Within the first 2 cycles of treatment, 12 weeks
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- ABlinatumomab 5/15/30 μg: Participants received blinatumomab by continuous intravenous infusion over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. The initial dose was 5 μg/m²/day for the first seven days of treatment, a dose of 15 μg/m²/day in the subsequent 7 days, followed by 30 μg/m²/day starting from Week 3 of treatment.
Arm/Group | Blinatumomab 15 μg | Blinatumomab 5/15 μg | ABlinatumomab 5/15/30 μg | Blinatumomab Overall
Number analyzed (Participants) | 7 | 23 | 6 | 36
percentage of participants | 14.3 [0.4 to 57.9] | 43.5 [23.2 to 65.5] | 66.7 [22.3 to 95.7] | 41.7 [25.5 to 59.2]

3. Secondary Outcome: Percentage of Participants With a Best Response of Complete Remission With Only Partial Hematological Recovery Within 2 Cycles of Treatment
Description: At the end of each infusion period, a bone marrow aspiration/biopsy was performed to evaluate the efficacy of blinatumomab. All hematological assessments of bone marrow were reviewed in a central reference laboratory. Complete remission with only partial hematological recovery (CRh*) was defined by the following criteria:
  * Less than or equal to 5% blasts in the bone marrow
  * No evidence of circulating blasts or extramedullar disease
  * Partial recovery of peripheral blood counts:
    * Platelets > 50,000/μL
    * Hemoglobin ≥ 7 g/dL
    * ANC > 500/μL.
Time Frame: Within the first 2 cycles of treatment, 12 weeks
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab 15 μg | Blinatumomab 5/15 μg | Blinatumomab 5/15/30 μg | Blinatumomab Overall
Number analyzed (Participants) | 7 | 23 | 6 | 36
percentage of participants | 57.1 [18.4 to 90.1] | 26.1 [10.2 to 48.4] | 0.0 [0.0 to 45.9] | 27.8 [14.2 to 45.2]

4. Secondary Outcome: Percentage of Participants With a Best Response of Partial Remission Within 2 Cycles of Treatment
Description: At the end of each infusion period, a bone marrow aspiration/biopsy was performed to evaluate the efficacy of blinatumomab. All hematological assessments of bone marrow were reviewed in a central reference laboratory. Partial remission was defined by the following criteria:
  • Bone marrow blasts ≤ 25%
Time Frame: Within the first 2 cycles of treatment, 12 weeks
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab 15 μg | Blinatumomab 5/15 μg | Blinatumomab 5/15/30 μg | Blinatumomab Overall
Number analyzed (Participants) | 7 | 23 | 6 | 36
percentage of participants | 0.0 [0.0 to 41.0] | 8.7 [1.1 to 28.0] | 0.0 [0.0 to 45.9] | 5.6 [0.7 to 18.7]

5. Secondary Outcome: Percentage of Participants With a Minimal Residual Disease (MRD) Response During the Core Study
Description: A minimal residual disease (MRD) response is defined as MRD < 10^-4 blasts/nucleated cells based on polymerase chain reaction (PCR) evaluation of individual rearrangements of immunoglobulin or T cell receptor genes.
Time Frame: During the core study treatment period (up to 30 weeks).
Population: Full analysis set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab 15 μg | Blinatumomab 5/15 μg | Blinatumomab 5/15/30 μg | Blinatumomab Overall
Number analyzed (Participants) | 7 | 23 | 6 | 36
percentage of participants | 71.4 [29.0 to 96.3] | 73.9 [51.6 to 89.8] | 50.0 [11.8 to 88.2] | 69.4 [51.9 to 83.7]

6. Secondary Outcome: Percentage of Participants Who Received an Allogeneic Hematopoietic Stem Cell Transplant (HSCT) After Treatment With Blinatumomab
Description: The percentage of participants who underwent immediate allogeneic HSCT (defined as those in remission who undergo HSCT without receiving any other treatments) after having discontinued or completed the core study.
Time Frame: Up to the data cut-off date of 15 October 2012; maximum follow up time was 459 days
Population: Full analysis set
Measure: Number; unit: percentage of participants
Groups:
- Blinatumomab: Participants received blinatumomab as a continuous intravenous infusion at a constant flow rate over 4 weeks followed by a 2-week treatment-free interval for up to 5 consecutive cycles.
Arm/Group | Blinatumomab 15 μg | Blinatumomab 5/15 μg | Blinatumomab 5/15/30 μg | Blinatumomab
Number analyzed (Participants) | 7 | 23 | 6 | 36
percentage of participants | 42.9 | 60.9 | 16.7 | 50.0

7. Secondary Outcome: Time to Hematological Relapse
Description: Time to hematological relapse was measured for participants who achieved a CR or CRh* during the core study and was measured from the time the participant first achieved remission until first documented relapse or death due to disease progression. Participants without a documented relapse (hematological or extramedullary) and who did not die were censored at the time of their last bone marrow assessment or their last survival follow-up visit confirming remission. Participants who died without having reported hematological relapse or without showing any clinical sign of disease progression were censored on their day of death.
  Hematological Relapse was defined as:
  * Proportion of blasts in bone marrow > 5%
  * Extramedullary relapse.
  Time to hematological relapse was analyzed by Kaplan-Meier methods.
Time Frame: Up to the data cut-off date of 15 October 2012; maximum follow up time was 459 days.
Population: Participants who reached complete remission or complete remission with partial hematological recovery during the core study.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Blinatumimab Overall: Participants received blinatumomab as a continuous intravenous infusion at a constant flow rate over 4 weeks followed by a 2-week treatment-free interval for up to 5 consecutive cycles.
Arm/Group | Blinatumomab 15 μg | Blinatumomab 5/15 μg | Blinatumomab 5/15/30 μg | Blinatumimab Overall
Number analyzed (Participants) | 5 | 16 | 4 | 25
days | 240.0 [63.0 to 270.0] | NA [227.0 to NA] — median was not reached during the core study | NA [15.0 to NA] — Median was not reached during the core study | 270.0 [227.0 to NA] — Could not be estimated due to the low number of events

8. Secondary Outcome: Relapse-free Survival
Description: Relapse-free survival was measured only for participants who achieved a CR or CRh* during the core study and was measured from the time the participant first achieved remission until first documented relapse or death due to any cause. Participants without a documented relapse (hematological or extramedullary) or who did not die were censored at the time of their last bone marrow assessment or their last survival follow-up visit confirming remission. Relapse-free survival was estimated using Kaplan-Meier methods.
Time Frame: Up to the data cut-off date of 15 October 2012; maximum follow up time was 459 days.
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Blinatumomab 15 μg | Blinatumomab 5/15 μg | Blinatumomab 5/15/30 μg | Blinatumomab Overall
Number analyzed (Participants) | 5 | 16 | 4 | 25
days | 137.0 [63.0 to 270.0] | 268.0 [226.0 to 403.0] | NA [15.0 to NA] — Median was not reached during the core study | 233.0 [175.0 to 291.0]

9. Secondary Outcome: Overall Survival
Description: Overall survival was measured for all participants from the date of first infusion of blinatumomab until the date of death due to any cause. Participants who did not die were censored on the last documented visit date. Overall survival was estimated using Kaplan-Meier methods.
Time Frame: Up to the data cut-off date of 15 October 2012; maximum follow up time was 667 days.
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Blinatumomab 15 μg | Blinatumomab 5/15 μg | Blinatumomab 5/15/30 μg | Blinatumomab Overall
Number analyzed (Participants) | 7 | 23 | 6 | 36
days | 269.0 [165.0 to 482.0] | 300.0 [254.0 to 431.0] | NA [276.0 to NA] — Median was not reached during the core study | 300.0 [258.0 to 455.0]

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Adverse events were evaluated for severity according to the grading scale provided in the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0 and according to the following:
  Grade I (mild); Grade 2 (moderate); Grade 3 (severe - significantly limits the patient's ability to perform routine activities despite symptomatic therapy; Grade 4 (life-threatening); Grade 5 (death).
  The investigator used medical judgment to determine if there was a causal relationship (ie, certain, probable, possible, unlikely, not related) between an adverse event and blinatumomab.
  A serious adverse event is any untoward medical occurrence or effect, that at any dose:
  resulted in death, was life-threatening, required or prolonged hospitalization, resulted in persistent or significant disability or incapacity, is a congenital anomaly or birth defect or is a medically important condition.
Time Frame: From the start of the first infusion to 30 days after the end of the last infusion in the core study or from the start of the first retreatment cycle infusion to 30 days after the end of the last retreatment cycle; median treatment duration was 55.7 days.
Population: Safety analysis set, defined as all participants who received any infusion of blinatumomab.
Measure: Number; unit: participants
Arm/Group | Blinatumomab 15 μg | Blinatumomab 5/15 μg | Blinatumomab 5/15/30 μg | Blinatumomab Overall
Number analyzed (Participants) | 7 | 23 | 6 | 36
participants
  Any adverse event (AE) | 7 | 23 | 6 | 36
  Adverse events of at least CTC grade 3 | 7 | 15 | 5 | 27
  Treatment-related adverse events | 7 | 23 | 6 | 36
  Related adverse events of at least CTC grade 3 | 7 | 12 | 4 | 23
  Serious adverse events | 6 | 13 | 5 | 24
  Serious adverse events of at least CTC grade 3 | 6 | 12 | 4 | 22
  Serious related adverse events | 4 | 8 | 4 | 16
  AEs leading to interruption of blinatumomab | 3 | 6 | 3 | 12
  AEs leading to discontinuation of blinatumomab | 4 | 4 | 1 | 9
  AEs leading to death | 1 | 4 | 1 | 6

11. Secondary Outcome: Steady State Blinatumomab Concentration
Description: The steady state concentration of blinatumomab was summarized as the observed concentrations collected at least 10 hours after the intravenous infusion was started for cycle 1 and cycle 2, respectively. Actual doses administered were used in the analysis.
  Concentrations below the limit of detection (3 pg/mL) were set to zero before data analysis and concentrations below the lower limit of quantitation (50 pg/mL) were excluded from analysis.
Time Frame: Samples were collected at predose and at 48 hours following start of infusion, when dose is escalated and on Days 8, 15, 22, and 29 of the first 2 cycles.
Population: Participants who received blinatumomab and who had available pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Blinatumomab 5 μg: Participants receiving blinatumomab 5 μg/m²/day.
- Blinatumomab 15 μg: Participants receiving blinatumomab 15 μg/m²/day.
- Blinatumomab 30 μg: Participants receiving blinatumomab 30 μg/m²/day.
Arm/Group | Blinatumomab 5 μg | Blinatumomab 15 μg | Blinatumomab 30 μg
Number analyzed (Participants) | 31 | 34 | 5
pg/mL | 167 (66) | 553 (238) | 1180 (820)

12. Secondary Outcome: Clearance of Blinatumomab
Description: Clearance was calculated as R0/Css; where R0 is the infusion rate (μg/m^2/hr) and Css is the steady state concentration.
Time Frame: as for outcome 11
Population: Participants who received blinatumomab and who had available pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: L/m^2/hr
Groups:
- Blinatumomab: All participants who received blinatumomab.
Arm/Group | Blinatumomab
Number analyzed (Participants) | 36
L/m^2/hr | 1.34 (0.61)

13. Secondary Outcome: Serum Cytokine Peak Levels
Description: The activation of immune effector cells was monitored by the measurement of peripheral blood cytokine levels including interleukin (IL)-2, IL-6, IL-10, tumor necrosis factor (TNF)-α and interferon gamma (IFN-γ) using multiplex cytometric bead assays. The lower limit of quantification (LLOQ) is 125 pg/mL and the limit of detection (LOD) is 20 pg/mL.
Time Frame: Samples were collected prior to treatment start (baseline), and at 2, 6, 24, and 48 hours after drug infusion start, and at these same time points when dose is escalated in each treatment cycle.
Population: Participants who received blinatumomab and who had evaluable pharmacodynamic data.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 36
pg/mL
  IL-6: Cycle 1 (N=35) | 2563 (5231)
  IL-6: Cycle 2 (N=22) | 212 (477)
  IL-6: Cycle 3 (N=11) | 21 (26)
  IL-10: Cycle 1 (N=35) | 1302 (2563)
  IL-10: Cycle 2 (N=22) | 351 (582)
  IL-10: Cycle 3 (N=11) | 419 (730)
  IFN-Ɣ: Cycle 1 (N=35) | 467 (1824)
  IFN-Ɣ: Cycle 2 (N=22) | 25 (28)
  IFN-Ɣ: Cycle 3 (N=11) | NA (NA) — Data below detection level of the assay
  IL-2: Cycle 1 (N=35) | 36 (49)
  IL-2: Cycle 2 (N=22) | NA (NA) — Data below detection level of the assay
  IL-2: Cycle 3 (N=11) | NA (NA) — Data below detection level of the assay
  TNF-α: Cycle 1 (N=35) | 60 (122)
  TNF-α: Cycle 2 (N=22) | NA (NA) — Data below detection level of the assay
  TNF-α: Cycle 3 (N=11) | NA (NA) — Data below detection level of the assay

ADVERSE EVENTS:
Time Frame: From the start of the first infusion to 30 days after the end of the last infusion in the core study or from the start of the first retreatment cycle infusion to 30 days after the end of the last retreatment cycle; median treatment duration was 55.7 days.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Blinatumomab Overall: All participants who received blinatumomab by continuous intravenous infusion during the core study.
Arm/Group | Blinatumomab 15 μg | Blinatumomab 5/15 μg | Blinatumomab 5/15/30 μg | Blinatumomab Overall
Serious Adverse Events (participants affected / at risk) | 6/7 | 13/23 | 5/6 | 24/36
Other Adverse Events (participants affected / at risk) | 7/7 | 23/23 | 6/6 | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab 15 μg (N=7) | Blinatumomab 5/15 μg (N=23) | Blinatumomab 5/15/30 μg (N=6) | Blinatumomab Overall (N=36)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Keratoconjunctivitis sicca (Eye disorders) | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 1 | 3
Cytokine release syndrome (Immune system disorders) | 1 | 1 | 1 | 3
Graft versus host disease (Immune system disorders) | 1 | 0 | 0 | 1
Candida sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Catheter site infection (Infections and infestations) | 3 | 1 | 0 | 4
Central nervous system infection (Infections and infestations) | 0 | 1 | 0 | 1
Febrile infection (Infections and infestations) | 1 | 0 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 2
Pneumonia fungal (Infections and infestations) | 0 | 1 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 2
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 1
C-reactive protein increased (Investigations) | 1 | 1 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 1 | 2
Dysgraphia (Nervous system disorders) | 0 | 1 | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 1 | 1 | 3
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 2 | 1 | 3
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab 15 μg (N=7) | Blinatumomab 5/15 μg (N=23) | Blinatumomab 5/15/30 μg (N=6) | Blinatumomab Overall (N=36)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 3 | 1 | 2 | 6
Lymphopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 3
Monocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 3 | 1 | 7
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 5 | 2 | 9
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2 | 2
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 2 | 2 | 0 | 4
Dry eye (Eye disorders) | 0 | 2 | 1 | 3
Eye pain (Eye disorders) | 1 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 1 | 1 | 0 | 2
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 1 | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 0 | 3
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 4 | 2 | 7
Diarrhoea (Gastrointestinal disorders) | 3 | 6 | 3 | 12
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Faecal incontinence (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 5 | 2 | 8
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2 | 5
Catheter site haematoma (General disorders) | 1 | 0 | 0 | 1
Catheter site haemorrhage (General disorders) | 0 | 0 | 1 | 1
Catheter site pain (General disorders) | 0 | 3 | 0 | 3
Chest pain (General disorders) | 2 | 3 | 0 | 5
Chills (General disorders) | 2 | 2 | 3 | 7
Fatigue (General disorders) | 5 | 8 | 5 | 18
General physical health deterioration (General disorders) | 0 | 2 | 0 | 2
Influenza like illness (General disorders) | 0 | 0 | 1 | 1
Localised oedema (General disorders) | 1 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 1 | 2
Mucosal inflammation (General disorders) | 1 | 2 | 1 | 4
Oedema peripheral (General disorders) | 6 | 5 | 3 | 14
Pyrexia (General disorders) | 5 | 18 | 6 | 29
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Acute graft versus host disease in skin (Immune system disorders) | 1 | 0 | 0 | 1
Adenovirus infection (Infections and infestations) | 0 | 0 | 1 | 1
Candidiasis (Infections and infestations) | 2 | 1 | 0 | 3
Cystitis (Infections and infestations) | 0 | 2 | 0 | 2
Cytomegalovirus chorioretinitis (Infections and infestations) | 0 | 0 | 1 | 1
Infection (Infections and infestations) | 1 | 1 | 1 | 3
JC virus infection (Infections and infestations) | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 4 | 1 | 6
Oral herpes (Infections and infestations) | 0 | 3 | 0 | 3
Otitis media (Infections and infestations) | 1 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 2 | 0 | 2
Pharyngitis (Infections and infestations) | 1 | 0 | 1 | 2
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 1 | 1 | 0 | 2
Sinusitis (Infections and infestations) | 2 | 0 | 1 | 3
Staphylococcal infection (Infections and infestations) | 1 | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 3
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1 | 1 | 4
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 1 | 5
Blood albumin decreased (Investigations) | 1 | 0 | 0 | 1
Blood amylase increased (Investigations) | 1 | 1 | 0 | 2
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 2
Blood calcium decreased (Investigations) | 1 | 0 | 0 | 1
Blood fibrinogen decreased (Investigations) | 1 | 0 | 0 | 1
Blood fibrinogen increased (Investigations) | 1 | 4 | 0 | 5
Blood immunoglobulin A decreased (Investigations) | 2 | 4 | 2 | 8
Blood immunoglobulin G decreased (Investigations) | 2 | 3 | 2 | 7
Blood immunoglobulin M decreased (Investigations) | 3 | 2 | 2 | 7
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 1 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 2 | 3 | 0 | 5
C-reactive protein increased (Investigations) | 3 | 5 | 1 | 9
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 1
Fibrin D dimer increased (Investigations) | 3 | 4 | 2 | 9
Gamma-glutamyltransferase increased (Investigations) | 4 | 3 | 0 | 7
Immunoglobulins decreased (Investigations) | 0 | 2 | 0 | 2
Lipase increased (Investigations) | 1 | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 2 | 1 | 0 | 3
Prothrombin time prolonged (Investigations) | 0 | 1 | 1 | 2
Reticulocyte count increased (Investigations) | 0 | 2 | 0 | 2
Vital capacity abnormal (Investigations) | 1 | 0 | 0 | 1
Weight decreased (Investigations) | 4 | 2 | 2 | 8
Weight increased (Investigations) | 3 | 7 | 3 | 13
pH urine decreased (Investigations) | 2 | 2 | 0 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 4
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 3
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0 | 5
Aphasia (Nervous system disorders) | 2 | 1 | 0 | 3
Apraxia (Nervous system disorders) | 1 | 1 | 0 | 2
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 4 | 0 | 5
Formication (Nervous system disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 2 | 11 | 4 | 17
Intention tremor (Nervous system disorders) | 1 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 2 | 1 | 3
Neurotoxicity (Nervous system disorders) | 0 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 3 | 0 | 4
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0 | 1
Tremor (Nervous system disorders) | 2 | 8 | 2 | 12
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 2
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 1
Fear (Psychiatric disorders) | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 2 | 0 | 3
Mental disorder due to a general medical condition (Psychiatric disorders) | 1 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 2 | 2 | 4
Incontinence (Renal and urinary disorders) | 1 | 0 | 1 | 2
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 1 | 1 | 0 | 2
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2 | 7
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 1 | 9
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 4
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 4
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 6 | 1 | 8
Rash generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2
Circulatory collapse (Vascular disorders) | 2 | 1 | 1 | 4
Flushing (Vascular disorders) | 1 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 2 | 5 | 1 | 8
Hypotension (Vascular disorders) | 3 | 0 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.